CLINICAL TRIAL: NCT01946048
Title: Safety and Efficacy Investigation of Patients With Ischemic Cardiomyopathy by Transplantation of Umbilical Cord Derived Mesenchymal Stem Cells
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Ischemic Cardiomyopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12276102D-Cardiac Disease
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cells (Experimental): Stem cells implantation Patients with severe coronary artery disease with ischemic cardiomyopathy managed with intramyocardial administration of allogeneic mesenchymal stem cells.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Procedure: Selected patients were randomly divided into a cell therapy group and a control group.
  Umbilical Cord Blood Derived Mesenchymal Stem Cells at a dose of 150-250 million.

SUMMARY:
The aim of the present study is to investigate safety and efficacy of intramyocardial implantation of allogeneic mesenchymal stem cells in patients with ischemic cardiomyopathy .

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a common disorder that can lead to heart failure. Not all people with CAD are eligible for today's standard treatments. One new treatment approach uses umbilical cord blood derived mesenchymal stem cells-specialized cells capable of developing into other types of cells-to stimulate growth of new blood vessels for the heart. The aim of the present study is to investigate safety and efficacy of intramyocardial implantation of allogeneic mesenchymal stem cells in patients with ischemic cardiomyopathy .

ELIGIBILITY:
Inclusion Criteria:

1. Age from 30 to 80 years
2. ischemic cardiomyopathy
3. Left ventricular infarction area seriously low movement to no movement
4. The low whole left ventricular systolic function (LVEF 45% or less)
5. Have line or quasi coronary interventional treatment
6. Willing to accept patients with follow-up evaluation
7. Have signed informed consent form approved by the ethics committee

Exclusion Criteria:

1. Non elevation between S-wave and T-wave in patients with acute myocardial infarction
2. No function damage in patients with acute myocardial infarction
3. Acute myocardial infarction complicated with left ventricular aneurysm intends to do surgery
4. Complications of acute myocardial infarction with other machines (including: ventricular septal perforation, papillary muscle rupture, etc.)
5. Acute infectious diseases
6. Blood system diseases, such as thrombocytopenia, severe anemia, leukemia, etc
7. Severe renal disease, creatinine clearance < 36 ml/min, serum creatinine > 265 umol/L
8. Laboratory tests suggest abnormal liver function, glutamate-pyruvate transaminase (ALT) > 4 times the upper limit of normal
9. Unstable cerebral lesions
10. malignant tumor
11. Cognitive dysfunction and dementia patients, patients with severe mental illness
12. Patients with severe physical disabilities can't regular follow-up
13. Other serious uncontrolled system disease
14. To prepare or have the pregnancy women patients
15. Have a percutaneous coronary intervention contraindications: high-risk patients, such as the digestive tract, and intracranial hemorrhage or contrast allergy
16. Cannot use the test dose atorvastatin
17. Is not completed in accordance with the requirements for test the timing of the magnetic resonance imaging (MRI), PET, SPECT, follow-up testing (e.g., patients with implanted pacemakers or artificial joint)
18. Patients unable or unwilling to sign a consent form

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The examination of heart function | Post cell transplantation: 1, 3, 6 months
  Left ventricular ejection fraction： Change in left ventricular ejection fraction assessed with echocardiography after intramyocardial implantation of allogeneic mesenchymal stem cells.

SECONDARY OUTCOMES:
all-cause mortality | Post cell transplantation: one year
all-cause morbidity | Post cell transplantation: one year
major adverse cardiac and cerebrovascular events | Post cell transplantation: one year

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — The First Hospital of Hebei Medical University; Gang Liu, Doctor, Study Director — The First Hospital of Hebei Medical University; Guoping Ma, Master, Principal Investigator — The First Hospital of Hebei Medical University; Jun Zhang, Master, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China